CLINICAL TRIAL: NCT06738524
Title: Effect of Digital Addiction on Orexin a Peptide and Sleep Quality
Brief Title: Digital Addiction, Sleep Quality and Orexin-A Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Zehra Incedal Sonkaya, Asst. Prof., Amasya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 182210
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Digital Addiction
Keywords: Digital addiction; Orexin-A; Sleep quality; Technology
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The research was conducted in two stages. In the first stage, the "Pittsburgh Sleep Quality Index" and "Digital Addiction Scale" were applied to all students. In the second stage, the experimental and control groups were created by analyzing the scores of the students from the Digital Addiction Scale for the intervention study. It was calculated with the power analysis that 42 participants should be included in the study. 21 participants were randomly assigned to the intervention group and 21 participants to the control group by lot. Blood samples were taken from the students assigned to the intervention and control groups before the training and their orexin-A levels were measured. Then, the digital addiction combating training program was applied to the intervention group. After the training program was completed, a post-test was applied to both groups and orexin-A levels were measured again.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Education (Experimental): The intervention group was given "Fighting with Digital Addiction" training.
  Interventions: Behavioral: Fighting with Digital Addiction

INTERVENTIONS:
Behavioral: Fighting with Digital Addiction — The purpose of this training is to raise awareness among young people about the signs, causes and consequences of addictive use of technology and how to avoid excessive use of technology and technology addiction.

SUMMARY:
This study aims to determine the level of digital addiction in university students where technology use is quite common, and to evaluate the relationship between digital addiction and orexin and sleep quality.

The main question it aims to answer is:

* Are digital addiction trainings given to students effective on digital addiction levels?
* Are digital addiction trainings given to students effective on sleep quality?
* Is there a relationship between digital addiction level and orexin-A peptide?

DETAILED DESCRIPTION:
The changes experienced in technology along with the developing world also bring about major changes in the lives of individuals. It is seen that technology is present in every aspect of life, especially the internet that enables widespread communication and the use of the tools and equipment developed accordingly is rapidly increasing especially in the young age group. It is stated that digital addiction is spreading very rapidly throughout the world and has many negative consequences on the daily life and health of the individual. Many health problems such as personality disorders, violence, increase in aggressive behavior, disruptions in the sleep-wake cycle, anxiety, and depression are associated with digital addiction. Orexins are hypothalamic neuropeptides that play a role in the regulation of many complex behaviors such as nutrition, sleep, and wakefulness. In recent studies, it is thought that orexin can cause behavioral addictions. Orexin plays a role in both the early and late stages of the addiction mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Individuals studying at Amasya University,
* Those who agree to participate in the study,
* Individuals who do not have any communication barriers

Exclusion Criteria:

* Individuals who are not students at Amasya University,
* Individuals with communication disabilities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Digital Addiction Scale | 4 weeks.
  A positive change in participants' digital addiction scores is expected at the end of the training program.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonkaya ZI, Yazgan B. The Effect of Digital Addiction Training on University Students' Digital Addiction, Sleep Quality, and Orexin-A Levels: Randomized Controlled Trial. BMC Psychol. 2025 Aug 12;13(1):903. doi: 10.1186/s40359-025-03247-1. PMID 40797228